CLINICAL TRIAL: NCT04227353
Title: Healthy Eating and Active Lifestyle After Bowel Cancer - HEAL ABC Workbook: Development and Feasibility Trial
Brief Title: Healthy Eating and Active Lifestyle After Bowel Cancer: HEAL ABC
Acronym: HEALABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jana Sremanakova, PhD student, Nutrition Research Assistant, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHS001653
Record Dates: First submitted 2019-12-09; First posted 2020-01-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer; Survivorship; Behavior, Health
Keywords: colorectal; cancer; diet; physical activity; survivorship; behaviour
MeSH Terms: conditions — Colorectal Neoplasms; Health Behavior; Neoplasms; Motor Activity; Behavior

STUDY DESIGN:
Intervention Model Description: The study is prospective randomised controlled trial, open label, exploratory/feasibility trial. The study aims to test the Healthy Eating and Active Lifestyle After Bowel Cancer - HEAL ABC intervention and HEAL ABC resources for feasibility and will inform a future definitive randomised controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEAL ABC (Experimental): Participants allocated to the intervention will be encouraged to follow the HEAL ABC resources in order to make a healthy eating and active lifestyle change. This will be achieved by setting specific goal(s) and by making concrete plan(s) to implement changes in their everyday life. Interventions will be delivered in the form of written resources that will guide participants. Supportive phone calls using motivational interviewing techniques will be provided to participants every two weeks to encourage lifestyle changes.
  Interventions: Behavioral: HEAL ABC
- HEALTH (No Intervention): Participants allocated to the control group will be referred to publicly available resources on healthy lifestyle recommendations but will not receive any additional support.

INTERVENTIONS:
Behavioral: HEAL ABC — Participants will be assigned their first booklet based on the one they perceive to be the easiest for setting an incremental goal and achieving it. After the participant achieves successful behaviour change, he or she can move more confidently to the next booklet. Support will be provided every two weeks over the phone for 12 weeks. During the follow-up period, participants will use the follow-up booklet which helps them to continue with changes they have made and encourage them to set new goals.
  Arms: HEAL ABC

SUMMARY:
Trial Design:

This is a feasibility randomised controlled trial.

Aim:

The study aims to test the Healthy Eating and Active Lifestyle After Bowel Cancer - HEAL ABC intervention and HEAL ABC resources for feasibility and will inform a future definitive randomised controlled trial (RCT).

Objectives:

1. Is it practical to run HEAL ABC study as a definitive randomised controlled trial?
2. Adherence to intervention, motivations, barriers and facilitators of CRC survivors to follow HEAL ABC.

Study Population:

Colorectal cancer survivors who completed surgery and/or active treatment.

Intervention:

The intervention group will use HEAL ABC resource with supportive telephone calls every two weeks during the intervention period and once a month during the follow up period.

Control:

Participants follow standard care recommendations.

Timing and duration:

3 months intervention with 6 months follow up period

DETAILED DESCRIPTION:
Background:

Investigators were awarded a grant to develop a lifestyle resource called HEAL ABC - the Healthy Eating and Active Lifestyle After Bowel Cancer. This resource is based on prevention guidelines of World Cancer Research Fund and American Institute of Cancer Research. The resource was developed in cooperation with a psychologist and so has incorporated behaviour change theory. Investigators organised focused groups with patients and healthcare professionals, and amended the resource based on their feedback.

In this study, investigators will test the HEAL ABC resource and the HEAL ABC intervention for its practicality before further studies will be conducted.

HEAL ABC consists of 10 booklets and supportive materials. The order for using the booklets is not specified. Participants will be assigned their first booklet based on the one they perceive to be the easiest for setting an incremental goal and achieving it. This means the participant starts with the booklet of the highest self-efficacy and after the participant achieves successful behaviour change, he or she can move more confidently to the next booklet. During the follow up period, participants will use the follow up booklet which helps them to continue with changes they have made and encourage them to set a new goals.

Participants in the intervention group will receive a supportive telephone call every two weeks during the intervention period (three months) and once a month during the six months follow up.

Participants allocated to the control group will given information about publicly available resources on healthy lifestyle recommendations. No additional support will be provided.

Primary Question/Objective:

Is it feasible to run a definitive RCT to determine the effectiveness of HEAL ABC? This study will address questions around suitability and practicality of using the HEAL ABC resource and the ability to run an intervention in relation to adherence, recruitment, retention rates and the ability to collect relevant data.

Secondary Question/Objective:

Adherence to intervention and the motivations, barriers and facilitators of CRC survivors to follow HEAL ABC.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥18
* Minimum 12 weeks post-surgery and/or active treatment
* Completed all active anti-cancer treatments, including surgery, radiotherapy or chemotherapy
* Body mass index ≥20 kg/m2 and no previous unintentional weight loss ≥5% of body weight in the previous six months.
* Identified as living an unhealthy lifestyle based on current recommendations - follow less than four of the WCRF/AICR recommendations on eligibility questionnaire
* Ability to work with computer, smart phone or tablet.
* Able to give informed consent.

Exclusion Criteria:

* Receiving treatment for malignancy.
* Secondary malignancy.
* Having short bowel syndrome, Crohn's disease, ulcerative colitis, diverticulitis or jejunostomy (due to requirement for a very specific diet).
* Previous stroke, congested cardiac failure or oedema.
* Hepatic or renal failure
* Less than 12 weeks post-surgery or active treatment.
* Meeting the requirements of a healthy lifestyle (follow four or more of the WCRF/AICR recommendations).
* Being on any therapeutic diets, multiple food intolerances or allergies.
* Unplanned weight loss of ≥10% in the previous 3-6 months.
* Cannot read or communicate in English (due to resource constraints of this PhD study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to intervention | 3 months
  Assessed as adherence to WCRF/AICR guidelines by using a scoring system for nutrition and physical activity guideline adherence developed by McCullough and colleagues. Number of goals set and number of changes implemented in everyday life during the 3 months intervention.
Adherence to intervention | 6 months
  Assessed as adherence to WCRF/AICR guidelines by using a scoring system for nutrition and physical activity guideline adherence developed by McCullough and colleagues. Number of goals set and number of changes implemented in everyday life during the 6 months follow up.
Recruitment rates | 3 months
  Cumulative recruitment against target rate each month.
Recruitment rates | 6 months
  Cumulative recruitment against target rate each month.
Retention rates | 3 months
  Calculated as the number of participants who completed the study divided by the number of participants randomised.
Retention rates | 6 months
  Calculated as the number of participants who completed the study divided by the number of participants randomised.
Acceptability of the intervention | 3 months
  This will be qualitatively assessed through in depth interviews with a subset of the trial participants.
Acceptability of the intervention | 6 months
  This will be qualitatively assessed through in depth interviews with a subset of the trial participants.
Data completion rates | 3 months
  Completeness of collected data will be assessed for all time points (% missing).
Data completion rates | 6 months
  Completeness of collected data will be assessed for all time points (% missing).

SECONDARY OUTCOMES:
Change in participants' experience, motivation, barriers and facilitators to use HEAL ABC resources and follow the intervention | 3 months and 6 months
  Qualitatively assessed with in depth interviews.
Change in behaviour | Baseline, 3 months and 6 months
  The health action process approach (HAPA) questionnaires, previously used in publications investigating changes in HAPA constructs in lifestyle interventions. A 5 point Likert scale will be used for each question. Minimum score is 15 and maximum score is 75. Higher score is better score.
Change in dietary intake | Baseline, 3 months and 6 months
  Three day dietary assessment. Participants will complete prospectively food diary during the day and enter all foods and drinks consumed into online system for dietary assessment - INTAKE24.
Change in BMI | Baseline, 3 months and 6 months
  Body weight [kg] and height [m] to calculate body mass index
Change in waist to hip ratio | Baseline, 3 months and 6 months
  waist circumference [cm] and hip circumference [cm] to calculate waist to hip ratio
Change in body composition (BIA) | Baseline, 3 months and 6 months
  lean mass [%] and fat mass [%] using bio-impedance machine
Change in body composition (CT scan) | Baseline, 3 months and 6 months
  muscle mass [cm2] and fat mass [cm2]using CT scans body composition analysis
Change in physical activity | Baseline, 3 months and 6 months
  Global Physical Activity Questionnaire is used to assess the metabolic equivalent (MET) based on Global Physical Activity Questionnaire Analysis Guide: https://www.who.int/ncds/surveillance/steps/resources/GPAQ_Analysis_Guide.pdf
Change in step count | Baseline, 3 months and 6 months
  pedometer
Patients' socio-demographic characteristics | Baseline
  age, gender, marital status, occupation, education, income, ethnicity, smoking status and number of supplements used
Contact with primary and secondary healthcare services | 6 months
  The Healthcare Resource Use Questionnaire - questionnaire was developed by a health economist for the EU funded project 'PreventIT' (2016-2018, grant number 689238) responding to the Horizon 2020, Personalised Health and Care call PHC-21: Advancing active and healthy aging with ICT: Early risk detection and intervention. There is no set score - questionnaire is used to estimate the costs associated with different healthcare services used.
Mortality | 6 months
  Patient's medical records
Morbidity | 6 months
  Patient's medical records
Change in Quality of life | Baseline, 3 months and 6 months
  SF-12 questionnaire - 12 questions, total score can range from 0 to 100 (sore zero indicates the lowest level of health and 100 indicates the highest level of health).

CONTACTS AND LOCATIONS:
Overall Officials: Jana Sremanakova, Principal Investigator — University of Manchester
Locations (3):
- United Kingdom (3):
  - Salford Royal NHS Foundation Trust, Manchester, Great Manchester
  - Manchester University NHS Foundation Trust, Manchester
  - The University of Manchester, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Investigators have published detailed study protocol and will share further details in main study publications
Supporting Information: Study Protocol
Time Frame: Study protocol has been published and is available online
Access Criteria: free access
URL: https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-020-00721-y

REFERENCES:
- [Background] Sremanakova J, Jones D, Cooke R, Burden S. Exploring Views of Healthcare Professionals, Researchers, and People Living with and beyond Colorectal Cancer on a Healthy-Eating and Active Lifestyle Resource. Nutrients. 2019 Oct 16;11(10):2482. doi: 10.3390/nu11102482. PMID 31623177
- [Background] Burden S, Jones DJ, Sremanakova J, Sowerbutts AM, Lal S, Pilling M, Todd C. Dietary interventions for adult cancer survivors. Cochrane Database Syst Rev. 2019 Nov 22;2019(11):CD011287. doi: 10.1002/14651858.CD011287.pub2. PMID 31755089
- [Background] Burden S, Sremanakova J, Jones D, Todd C. Dietary interventions for cancer survivors. Proc Nutr Soc. 2019 Feb;78(1):135-145. doi: 10.1017/S0029665118002690. Epub 2018 Dec 19. PMID 30563580
- [Background] Wright SJ, Gibson D, Eden M, Lal S, Todd C, Ness A, Burden S. What are colorectal cancer survivors' preferences for dietary advice? A best-worst discrete choice experiment. J Cancer Surviv. 2017 Dec;11(6):782-790. doi: 10.1007/s11764-017-0615-2. Epub 2017 Apr 20. PMID 28429186
- [Background] Aubrey V, Hon Y, Shaw C, Burden S. Healthy eating interventions in adults living with and beyond colorectal cancer: a systematic review. J Hum Nutr Diet. 2019 Aug;32(4):501-511. doi: 10.1111/jhn.12651. Epub 2019 Apr 3. PMID 30941834
- [Derived] Sremanakova J, Sowerbutts AM, Todd C, Cooke R, Burden S. Healthy Eating and Active Lifestyle After Bowel Cancer (HEAL ABC): feasibility randomised controlled trial protocol. Pilot Feasibility Stud. 2020 Nov 13;6(1):176. doi: 10.1186/s40814-020-00721-y. PMID 33292854